CLINICAL TRIAL: NCT06744582
Title: Estimating VO2 Max and Recovery in Patients Undergoing Total Hip Arthroplasty: A Feasibility Study
Brief Title: Estimating VO2 Max and Recovery
Status: Recruiting | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Nuffield Health Bournemouth (Unknown)
Responsible Party: Principal Investigator, Tom Wainwright, Professor of Orthopaedics, Bournemouth University
Other Study IDs: ORI/VO2/24
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hip Osteoarthritis
Keywords: Osteoarthritis; Hip arthroplasty; Hip replacement; Musculoskeletal; VO2 max; Cardiovascular fitness
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VO2 max — The aim of this study is to generate data on the estimation of natural variation in VO2 max changes before and after surgery using seismocardiography.

SUMMARY:
The study aims to estimate VO2 max levels at pre- and post-operative timepoints before and after hip arthroplasty surgery, using non-exercise-based measurement methods.

DETAILED DESCRIPTION:
This observational cohort study will measure an estimation of VO2 max prior to and following routine robotic arm assisted hip arthroplasty surgery, and examine its association with outcomes of recovery after surgery. Although VO2 max is usually measured using cardiopulmonary exercise testing, these tests are often unachievable for an elderly population with end stage hip osteoarthritis and in a lot of pain. For this reason, this study will estimate VO2 max using the Seismofit® System. This works by measuring vibrations arising from heart beats that are transmitted to the chest. The small Seismofit® device is battery powered, and uses Bluetooth to communicate the results to a smartphone app. The device is simply attached to the lower part of the participant's sternum using an adhesive patch and takes around 45 seconds to record the data.

The study will also assess recovery through measuring pain and functional ability via patient reported outcome measures (PROMs) and objective performance assessments. In addition, participants will be invited to wear activity monitors on their wrist prior to surgery, and for 12 weeks after surgery, to understand changes in physical activity and sleep patterns.

Patients undergoing a robot-assisted hip arthroplasty with Professor Middleton at the Nuffield Health Hospital will be invited to take part in the study by the clinical team at Nuffield, and will be given a patient information sheet. If they are interested in taking part in the study, they will be contacted by a member of the research team at BU and invited into ORI to give their informed consent. Once the participant has consented, they will undergo pre-surgery assessments. It is anticipated that it will take 12 months to recruit the 30 participants. Participants will then have follow-up study visits on Day-1 at Nuffield Hospital, and at 3-, 6-, and 12-weeks post-surgery at ORI. Data relating to surgery, discharge and medication will also be taken from routine data collected at Nuffield Hospital. Participants will continue to be followed up clinically as per standard care at Nuffield Hospital. Findings from this feasibility study will inform the design of future interventions to improve cardiovascular fitness in patients undergoing hip arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years;
* Undergoing total hip replacement at Nuffield Hospital;
* Voluntary written Informed Consent obtained;
* Participant able to complete study follow-up.

Exclusion Criteria:

* Requiring revision hip arthroplasty;
* Patients with implanted electronic equipment, such as a pacemaker;
* Women judged by the Investigator to be of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period;
* Unable to provide informed consent (insufficient English, lives overseas, unable to return easily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Robot Assisted Total Hip Replacement at the Nuffield Health
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Natural variation in VO2 max | From enrollment to 12 weeks after surgery
  VO2 max will be estimated using seismocardiography prior to surgery, on day 1, and at 3 weeks, 6 weeks, and 12 weeks following surgery.

SECONDARY OUTCOMES:
Patient Reported Outcome Measure (PROM) - The Hip Disability and Osteoarthritis Outcome Score (HOOS) | From enrollment to 12 weeks after surgery
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) will be assessed at pre-surgery, 3 weeks, 6 weeks, and 12 weeks following surgery. There are 5 subscales (pain, symptoms and stiffness, activities of daily living, function in sports and recreational activities, and quality of life), that are all scored individually on a scale of 0 to 100, with 0 indicating extreme symptoms and 100 indicating no symptoms.
Functional Assessment - 30 Second Chair Stand Test | From enrollment to 12 weeks after surgery
  30s Chair Stand Test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6 weeks, and 12 weeks following surgery.
Functional Assessment - 40 Metre Fast-Paced Walk Test | From enrollment to 12 weeks after surgery
  40m Fast-Paced Walk Test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6 weeks, and 12 weeks following surgery.
Functional Assessment - Stair Climb Test | From enrollment to 12 weeks after surgery
  Stair Climb Test as recommended by the Osteoarthritis Research Society International (OARSI). Assessment will be done prior to surgery, and again at 3 weeks, 6 weeks, and 12 weeks following surgery.
Monitoring of physical activity | From enrollment to 12 weeks after surgery
  Participants will be invited to wear an activity monitor on their wrist for at least three consecutive days prior to surgery, and for the 12 weeks following discharge. The Actiwatch device is a wrist-worn activity data recorder that records the amount of physical activity the patient does by measuring the motion in the wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Wainwright, Principal Investigator — Bournemouth University
Locations (2):
- United Kingdom (2):
  - Nuffield Health Hospital Bournemouth, Bournemouth, Dorset
  - Bournemouth University, Bournemouth, Dorset

IPD SHARING:
Plan to Share IPD: No